CLINICAL TRIAL: NCT05597956
Title: Effectiveness of Infiltration Resins in the Treatment of Enamel Defects in Child Patients
Brief Title: Effectiveness of Infiltration With Resin in Treatment of MIH Incisors in Children Showing Opacities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Montserrat Catalá Pizarro, Associate Professor, University of Valencia
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: O00017836e2200003229
Record Dates: First submitted 2022-10-20; First posted 2022-10-28 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Children, Adult; Molar Incisor Hypomineralization; Dental Diseases; Opacity; Anterior Teeth
MeSH Terms: conditions — Molar Hypomineralization; Stomatognathic Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- white defects (Experimental): Evaluate the infiltration of the defects.
  Interventions: Procedure: yellow defects; Procedure: brown defects
- yellow defects (Experimental): Evaluate the infiltration of the defects.
  Interventions: Procedure: white defects; Procedure: brown defects
- Brown defects (Experimental): Evaluate the infiltration of the defects.
  Interventions: Procedure: white defects; Procedure: yellow defects

INTERVENTIONS:
Procedure: white defects — "With the previously cleaned tooth, the enamel will be prepared with a product that makes it more porous, thus eliminating the decalcified areas of the deepest part of the lesion. After completely removing the water from the surface, the resin will be applied infiltrating between the canaliculi of the enamel. When polymerized, it will form a framework that will seal the surface, thus improving surface resistance and aesthetics by modifying the refractive indices of the affected enamel, mimicking it with the remaining healthy enamel".
  Arms: Brown defects; yellow defects
Procedure: yellow defects — "With the previously cleaned tooth, the enamel will be prepared with a product that makes it more porous, thus eliminating the decalcified areas of the deepest part of the lesion. After completely removing the water from the surface, the resin will be applied infiltrating between the canaliculi of the enamel. When polymerized, it will form a framework that will seal the surface, thus improving surface resistance and aesthetics by modifying the refractive indices of the affected enamel, mimicking it with the remaining healthy enamel".
  Arms: Brown defects; white defects
Procedure: brown defects — "With the previously cleaned tooth, the enamel will be prepared with a product that makes it more porous, thus eliminating the decalcified areas of the deepest part of the lesion. After completely removing the water from the surface, the resin will be applied infiltrating between the canaliculi of the enamel. When polymerized, it will form a framework that will seal the surface, thus improving surface resistance and aesthetics by modifying the refractive indices of the affected enamel, mimicking it with the remaining healthy enamel".
  Arms: white defects; yellow defects

SUMMARY:
Enamel development defects are the result of a set of environmental, systemic and genetic causal agents that reveal a multifactorial etiology model, which in anterior teeth produces a serious aesthetic problem, converted into a problem of visual perception. In hypomineralized enamel, light rays encounter multiple interfaces between organic and mineral fluids, with different refractive indices. At each interface, the light is deflected and reflected, producing an overexposed "optical labyrinth" that is perceived as a yellow, white, or brown stain.

The term "infiltration" has been modified and developed commercially in Germany for the treatment of non-cavitated caries on smooth and proximal surfaces, in which the porosities of the enamel lesion are infiltrated with a low-viscosity resin, thus creating a barrier of diffusion, without the need for any type of additional material on the tooth surface.

An added positive effect of infiltration with the queens is that the enamel lesions lose their whitish appearance when the microporosities are filled, mimicking the area of the lesion with the remaining healthy enamel. This effect is what has led clinicians to adapt this treatment for the management of enamel defects.

Given the growing interest in the treatment of opacities in the anterior sector, due to the demanding contemporary aesthetic requirements, and the increased acceptance of minimally invasive therapies, the need has been seen to seek greater predictability for the treatment of defects. of conservative enamel from an early age and offer effective therapeutic alternatives.

ELIGIBILITY:
Inclusion Criteria:

. Pediatric patients, aged between 9 and 16 years.

* Patients who have molar incisor hypomineralization, any lesion with isolated opacities or discoloration of the permanent incisors.
* Patients who present at least one opacity in the central incisors.
* Go to the dental clinic for revision or treatment of the University of Valencia.

Exclusion Criteria:

* Opacities with loss of enamel or tooth structure, active caries lesions, clinical symptoms of irreversible pulpitis such as spontaneous pain or persistent pain, a history of using bleaching agents, with intolerance to any milk protein, who have an allergic pathology or syndromic or uncooperative during the clinical procedure.

Ages: 9 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2023-09-19 (Actual); Primary Completion 2024-09-12 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Change in the color of opacities | Between five and six months
  Measured in color changes of opacities using the CIE L*A*B* system. The color of (coated) objects is visualized and quantified by using the CIELAB color space. The 3-dimensional color space is built-up from three axes that are perpendicular to one another.The L*-axis gives the lightness: a white object has an L* value of 100 and the L* value of a black object is 0. The so-called achromatic colors, the shades of grey, are on the L*-axis.
  Chromatic ('real') colors are described by using the two axes in the horizontal plane. The a*-axis is the green-red axis and the b*-axis goes from blue (-b*) to yellow (+b*).its measurement is possible thanks to the spectrophotometer.
  Clinical improvement and better visual perception of infiltrated enamel defects
Change in the density of opacities | Between five and six months
  DIAGNOdent is a diagnostic method based on an intermittent red fluorescence laser with a wavelength of 655 nm and 1 mW (milliwatt )that penetrates several millimeters from the tooth surface.

SECONDARY OUTCOMES:
aesthetic change of opacities | Between five and six months
  Satisfaction questionnaire. A post-treatment questionnaire will be passed with questions regarding the satisfaction of the patient and parents. The results will be classified from 0 to 4, with 0 being not at all satisfied and 4 being very satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No
The project will be carried out by a research team. Where there will be a principal investigator, and a collaborator who will carry out the clinical experimentation part.

REFERENCES:
- [Derived] Casana-Ruiz MD, Vello-Ribes MA, Catala-Pizarro M. Resin Infiltration for Anterior Teeth Affected by Molar Incisor Hypomineralization in Children and Adolescents: A Clinical Study of Color Masking, Sensitivity, and Aesthetic Perception: A Prospective Single-Arm Interventional Clinical Study. Children (Basel). 2026 Jan 15;13(1):131. doi: 10.3390/children13010131. PMID 41597140